CLINICAL TRIAL: NCT00191646
Title: Phase III Randomized Trial of Induction Chemotherapy With Gemcitabine and Carboplatin Followed by Elective Paclitaxel Consolidation Versus Paclitaxel and Carboplatin Followed by Elective Paclitaxel Consolidation in Patients With Primary Epithelial Ovarian, Primary Peritoneal Cancer or Fallopian Tube Carcinoma
Brief Title: An Ovarian, Primary Peritoneal or Fallopian Tube Cancer Study for Patients That Have Not Received Prior Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6891; B9E-US-S302 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Results first posted 2010-09-09 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-02

CONDITIONS: Genital Neoplasms, Female; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pelvic Neoplasms; Peritoneal Neoplasms
MeSH Terms: conditions — Genital Neoplasms, Female; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pelvic Neoplasms; Peritoneal Neoplasms | interventions — Gemcitabine; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine/Carboplatin (Experimental): Gemcitabine 1000 milligrams per meter square (mg/m^2) Day 1 and Day 8, Carboplatin Area Under the Curve (AUC) 5 Day 1, six 21-day cycles
  Interventions: Drug: Gemcitabine; Drug: Carboplatin
- Paclitaxel/Carboplatin (Active Comparator): Paclitaxel 175 milligrams per meter square (mg/m^2) administered intravenously (IV) Day 1 Carboplatin AUC 6 Day 1, six 21 day cycles
  Interventions: Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Gemcitabine — 1000 mg/m^2, Intravenously (IV), day 1 and day 8 every (q) 21 days x 6 cycles
  If anything other than complete response in Paclitaxel arm patients, 1000 mg/m^2, IV, day 1 and day 8 q 21 days until complete response, disease progression or unacceptable toxicity
  Other Names: LY188011; Gemzar
  Arms: Gemcitabine/Carboplatin
Drug: Paclitaxel — 175 mg/m^2, IV, Day 1, q 21 days x 6 cycles
  If complete response both Paclitaxel and Gemcitabine arms may elect to receive consolidation therapy, 135 mg/m^2, IV, 3 hours q 28 days x 12 cycles (1 year)
  If no complete response, then Gemcitabine arm patients may receive 175 mg/m^2, IV, Day 1, q 21 days until complete response, disease progression or unacceptable toxicity
  Arms: Paclitaxel/Carboplatin
Drug: Carboplatin — Gemcitabine/Carboplatin AUC 5, IV, Day 1, q 21 days x 6 cycles
  Paclitaxel/Carboplatin AUC 6, IV, Day 1, q 21 days x 6 cycles

SUMMARY:
This is a phase III randomized study comparing induction treatments of Gemcitabine and Carboplatin versus Paclitaxel and Carboplatin, with or without consolidation therapy for patients that do not have any evidence of disease after completion of six cycles of induction therapy. Patients with disease after induction therapy will crossover to receive single agent therapy.

DETAILED DESCRIPTION:
This study (Study B9E-US-S302) is a multicenter, comparative, open-label randomized, superiority, trial evaluating Gemcitabine and Carboplatin to the standard of care. Both treatment arms will be given the option to receive elective consolidation therapy of Paclitaxel 135 mg/m^2 given every 28 days for one year. Patients not achieving a complete response will crossover to the opposite single agent.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with a histologic diagnosis of primary peritoneal carcinoma, epithelial ovarian carcinoma or fallopian tube carcinoma Stage IC, II, III or IV.
* All patients must have had surgery for fallopian, ovarian or peritoneal carcinoma to establish the diagnosis and have tissue available for histologic evaluation and confirmation of organ of origin.
* Patients must be enrolled no more than twelve weeks postoperatively.
* Patients must be willing to receive their chemotherapy drugs intravenously, as intraperitoneal therapy is not part of this trial.

Key Exclusion Criteria:

* Patients with a current diagnosis of epithelial ovarian tumor of low malignant potential (Borderline carcinomas) are not eligible.
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis are excluded
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor are excluded
* With the exception of non-melanoma skin cancer and other specific malignancies patients who had (or have) any evidence of the other cancer present within the last 5 years or whose previous cancer treatment contraindicates this protocol therapy are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2002-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) OR 1-317-615-4559 MON-FRI 9AM -5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (55):
- United States (54):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Gatos, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Modesto, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Englewood, Colorado
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newark, Delaware
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Myers, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sunrise, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Savannah, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palatine, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Indianapolis, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., South Bend, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Metairie, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scarborough, Maine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Detroit, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Duluth, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minneapolis, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St Louis, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Billings, Montana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Las Vegas, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reno, Nevada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hackensack, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chapel Hill, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dayton, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dunmore, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Johnstown, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sayre, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Providence, Rhode Island
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chattanooga, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Knoxville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lubbock, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Roanoke, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madison, Wisconsin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 919 patients were randomized, only 831 randomized patients were included in any analyses. 85 randomized patients were excluded due to significant noncompliant issues and 3 patients were excluded due to unavailable data.
Groups:
- Gemcitabine/Carboplatin: Induction: Gemcitabine 1000 mg/m^2 Days 1 and 8 followed by Carboplatin Area Under the Curve (AUC) 5 Day 1; every 21-days.
  Consolidation (gemcitabine to paclitaxel): Paclitaxel 135 mg/m^2 Intravenous Piggy-Back (IVPB), 3 hours every 28 days for 12 cycles (one year).
  Paclitaxel (crossover): Single agent Paclitaxel 175 mg/m^2 day 1 to be repeated every 21 days.
- Paclitaxel/Carboplatin: Induction: Paclitaxel 175 mg/m^2 and Carboplatin AUC 6 Day 1, every 21 days. Consolidation (paclitaxel to paclitaxel): Paclitaxel 135 mg/m^2 IVPB, 3 hours every 28 days for 12 cycles (one year).
  Gemcitabine (crossover): Single agent Gemcitabine 1000 mg/m^2 days 1, 8 to be repeated every 21 days.
Period: Overall Study
Arm/Group | Gemcitabine/Carboplatin | Paclitaxel/Carboplatin
Started | 417 | 414
Received Induction Therapy | 411 | 409
Received Consolidation Therapy | 169 | 183
Received Crossover Therapy | 77 | 78
Completed | 246 (Completed was defined as the patients treated in either consolidation therapy or crossover therapy.) | 261 (Completed was defined as the patients treated in either consolidation therapy or crossover therapy.)
Not Completed | 171 | 153
Not completed — Toxicity | 26 | 37
Not completed — Disease Progression | 5 | 6
Not completed — Physician Decision | 20 | 11
Not completed — Withdrawal by Subject | 58 | 39
Not completed — Protocol Violation | 5 | 7
Not completed — Death | 6 | 8
Not completed — Other | 33 | 34
Not completed — Missing Data | 18 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gemcitabine/Carboplatin | Paclitaxel/Carboplatin | Total
Number analyzed (Participants) | 417 | 414 | 831
Age Continuous [Mean (Standard Deviation); unit: years] | 59.7 (11.4) | 60.3 (10.8) | 60.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 417 | 414 | 831
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 379 | 379 | 758
  Black or African American | 12 | 13 | 25
  Asian | 5 | 5 | 10
  Native American | 2 | 1 | 3
  Other | 19 | 16 | 35
Organ of Origin [Number; unit: participants] — Organ from which disease originated
  participants
    Ovary | 355 | 362 | 717
    Peritoneum | 56 | 50 | 106
    Missing Data | 6 | 2 | 8
Extent of Residual Disease [Number; unit: participants] — Patients either had no clinical evidence of residual disease (non-measurable), either by physical or radiologic exam, that was measurable as defined below or they had residual disease that was measured by either of the following techniques. Measurable lesions were those which could be measured accurately and followed in at least one dimension (the longest dimension being the one recorded). Each lesion must be >= 20 millimeters (mm) when measured by conventional techniques [palpation, plain X-ray, Computed tomography (CT), and Magnetic resonance imaging (MRI)], or >= 10 mm by spiral CT.
  participants
    Measurable | 139 | 114 | 253
    Non-measurable | 276 | 300 | 576
    Missing Data | 2 | 0 | 2
Zubrod Performance Status [Number; unit: participants] — 0 Asymptomatic
  1. Symptomatic, fully ambulatory
  2. Symptomatic, in bed < 50% of the day
  3. Symptomatic, in bed > 50% of the day but not bedridden
  4. Bedridden
  5. Dead
  participants
    0 | 239 | 232 | 471
    1 | 139 | 157 | 296
    2 | 27 | 16 | 43
    >= 3 | 0 | 0 | 0
    Missing Data | 12 | 9 | 21
International Federation of Gynecology and Obstetrics (FIGO) Stage at Initial Surgery [Number; unit: participants] — Ic: Tumor is either Stage IA or IB level but the capsule is ruptured or there is tumor on the ovarian surface or malignant cells are present in ascites or washings.
  II: Tumor involves one or both ovaries with pelvic extension
  III: Tumor involving one or both ovaries, with microscopically confirmed peritoneal metastases outside the pelvis and/or regional lymph node metastases
  IV: Distant metastases (Excludes peritoneal metastases)
  participants
    Stage Ic | 21 | 22 | 43
    Stage II | 44 | 39 | 83
    Stage III | 284 | 289 | 573
    Stage IV | 68 | 63 | 131
    Missing Data | 0 | 1 | 1
Histology [Number; unit: participants]
  Mucinous | 10 | 10 | 20
  Serous | 283 | 276 | 559
  Endometroid | 44 | 40 | 84
  Undifferentiated | 7 | 7 | 14
  Clear Cell | 21 | 23 | 44
  Mixed Epithelial | 9 | 13 | 22
  Transitional Cell | 3 | 1 | 4
  Malignant Brenner's Tumor | 0 | 0 | 0
  Adenocarcinoma Not Otherwise Specified (NOS) | 22 | 23 | 45
  Other | 17 | 21 | 38
  Missing Data | 1 | 0 | 1
Volume of Residual Tumor Following Debulking Surgery [Number; unit: participants]
  < 2 centimeters | 309 | 314 | 623
  >= 2 centimeters | 102 | 96 | 198
  Missing Data | 6 | 4 | 10
CA-125 Units per milliliter at Baseline for All Patients [Mean (Standard Deviation); unit: units per milliliter] — Cancer Antigen 125, units per milliliter
  units per milliliter | 492.772 (1138.556) | 479.854 (1117.040) | 486.329 (1127.213)

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival was defined as the duration from the date of randomization to the first date of documented disease progression or death from any cause. Tumor assessments were performed every three 21-day cycles during induction and crossover. Progression free survival was censored at the date of the last follow-up visit for participants who were still alive and who had not progressed. Results are presented as a comparison between the two study treatment sequences (induction therapy followed by elective consolidation or crossover therapy) rather than the two induction therapies.
Time Frame: Baseline to measured progressive disease or death up to 82 months
Population: Intent to treat (ITT) population, which includes all randomized participants. 3 participants in the Gemcitabine/Carboplatin treatment sequence were excluded due to missing data, and 1 participant in the Paclitaxel/Carboplatin treatment sequence was excluded for missing data. G/C Arm: 292 events, 122 censored. P/C Arm: 279 events, 134 censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gemcitabine/Carboplatin | Paclitaxel/Carboplatin
Number analyzed (Participants) | 414 | 413
Months | 20.0 [17.9 to 22.2] | 22.2 [19.0 to 25.7]
Statistical Analysis 1: Comparison: Gemcitabine/Carboplatin vs Paclitaxel/Carboplatin; Using a two-sided log-rank test with a Type I error of 0.05, 636 events for PFS out of the 919 patients would give an 80% statistical power under the alternative hypothesis that the hazard ratio of the G/C arm versus the P/C arm was 0.08; Test type: Superiority or Other; p = 0.199, Log Rank

2. Secondary Outcome: Proportion of Participants With Response (Response Rate)
Description: Response rate (RR) = proportion of participants with best overall Complete Response (CR: disappearance of all target lesions [TL]) or Partial Response (PR: 30% decrease in sum of longest diameter of TL). Induction therapy RR = number of participants with CR or PR during induction divided by number of participants with measurable disease at baseline (TL measurement during screening). Crossover therapy RR = number of participants with CR or PR during crossover divided by number of participants with measurable disease at baseline (latest TL measurement by first dose date of crossover therapy).
Time Frame: Baseline to measured progressive disease up to 82 months
Population: All ITT participants with measurable disease at baseline (screening) for induction period; all ITT participants who crossed over to single agent therapy and had measurable disease before or at crossover for crossover period. Participants in consolidation therapy achieved CR during induction therapy and were not included in analysis.
Measure: Mean (95% Confidence Interval); unit: proportion of responders
Groups:
- Gemcitabine/Carboplatin (Induction): Gemcitabine 1000 milligrams per meter square (mg/m^2) Day 1, Day 8, Carboplatin AUC 5 Day 1, six 21-day cycles
- Paclitaxel/Carboplatin (Induction): Paclitaxel 175 milligrams per meter square (mg/m^2) administered intravenously (IV) Day 1 Carboplatin AUC 6 Day 1, six 21-day cycles
- Gemcitabine (Crossover): Crossover (From Paclitaxel to Gemcitabine) - If no complete response on Paclitaxel, patient crossed over to receive Gemcitabine 1000 mg/m^2, IV, day 1 and day 8 q 21 days until complete response, disease progression or unacceptable toxicity
- Paclitaxel (Crossover): Crossover (From Gemcitabine to Paclitaxel) - If no complete response on Gemcitabine, patient crossed over to receive Paclitaxel 175 mg/m^2, IV, day 1, q 21 days until complete response, disease progression or unacceptable toxicity
Arm/Group | Gemcitabine/Carboplatin (Induction) | Paclitaxel/Carboplatin (Induction) | Gemcitabine (Crossover) | Paclitaxel (Crossover)
Number analyzed (Participants) | 139 | 114 | 28 | 33
proportion of responders | 0.676 [0.638 to 0.798] | 0.711 [0.651 to 0.822] | 0.357 [0.194 to 0.576] | 0.303 [0.161 to 0.500]
Statistical Analysis 1: Comparison: Gemcitabine/Carboplatin (Induction) vs Paclitaxel/Carboplatin (Induction); Test type: Superiority or Other; p = 0.771, Fisher Exact
Statistical Analysis 2: Comparison: Gemcitabine (Crossover) vs Paclitaxel (Crossover); Test type: Superiority or Other; p = 0.784, Fisher Exact

3. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure was defined as the duration from date of randomization to the date of the first of the following events: early discontinuation of study therapy; progression of disease, or death due to any cause. Time to treatment failure will be censored at the date of the last follow-up visit for participants who did not discontinue early, who are still alive, and who have not progressed. Results are presented as a comparison between the two study treatment sequences (induction therapy followed by elective consolidation or crossover therapy) rather than the two induction therapies.
Time Frame: Baseline to stopping treatment up to 82 months
Population: Intent to treat (ITT) population, which includes all randomized participants. 3 participants in the Gemcitabine/Carboplatin treatment sequence were excluded due to missing data, and 1 participant in the Paclitaxel/Carboplatin treatment sequence was excluded for missing data. G/C Arm: 336 events, 78 censored. P/C Arm: 330 events, 83 censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Carboplatin | Paclitaxel/Carboplatin
Number analyzed (Participants) | 414 | 413
months | 13.0 [11.7 to 15.1] | 13.1 [11.4 to 14.3]
Statistical Analysis 1: Comparison: Gemcitabine/Carboplatin vs Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.621, Log Rank

4. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the duration from baseline to death. For participants who are still alive at the data cut-off date, survival will be censored at the last contact date. Results are presented as a comparison between the two study treatment sequences (induction therapy followed by elective consolidation or crossover therapy) rather than the two induction therapies.
Time Frame: Baseline to death from any cause up to 82 months
Population: Intent to treat (ITT) population, which includes all randomized participants. 3 participants in the Gemcitabine/Carboplatin treatment sequence were excluded due to missing data, and 1 participant in the Paclitaxel/Carboplatin treatment sequence was excluded for missing data. G/C Arm: 194 events, 220 censored. P/C Arm: 159 events, 254 censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine/Carboplatin | Paclitaxel/Carboplatin
Number analyzed (Participants) | 414 | 413
months | 43.8 [38.8 to 48.4] | 57.3 [48.5 to 64.0]
Statistical Analysis 1: Comparison: Gemcitabine/Carboplatin vs Paclitaxel/Carboplatin; Test type: Superiority or Other; p = 0.013, Log Rank

ADVERSE EVENTS:
Description: A participant was randomized to P/C but treated with G/C, and thus included in the P/C arm ITT population (disposition and efficacy tables) and included in the G/C arm of treated population (AE tables). This results in an inconsistency between number of participants analyzed and participant flow module.
Groups:
- Gemcitabine/Carboplatin Induction: Gemcitabine 1000 milligrams per meter square (mg/m2) Day 1, Day 8, Carboplatin AUC 5 Day 1, 6 21 day cycles
- Paclitaxel/Carboplatin Induction: Paclitaxel 175 milligrams per meter square (mg/m2) administered intravenously (IV) Day 1 Carboplatin AUC 6 Day 1, 6 21 day cycles
- Consolidation (Gemcitabine to Paclitaxel); Consolidation (Paclitaxel to Paclitaxel): Paclitaxel 135mg/m2 IV/3 hours every 28 days for 12 cycles (one year).
- Crossover (Paclitaxel to Gemcitabine): Single agent Gemcitabine 1000mg/m2 IV, Day 1, Day 8 to be repeated every 21 days.
- Crossover (Gemcitabine to Paclitaxel): Single agent Paclitaxel 175mg/m2 IV Day 1 to be repeated every 21 days.
Arm/Group | Gemcitabine/Carboplatin Induction | Paclitaxel/Carboplatin Induction | Consolidation (Gemcitabine to Paclitaxel) | Consolidation (Paclitaxel to Paclitaxel) | Crossover (Paclitaxel to Gemcitabine) | Crossover (Gemcitabine to Paclitaxel)
Serious Adverse Events (participants affected / at risk) | 96/412 | 72/408 | 14/169 | 12/183 | 8/78 | 8/77
Other Adverse Events (participants affected / at risk) | 404/412 | 394/408 | 157/169 | 170/183 | 76/78 | 73/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Carboplatin Induction (N=412) | Paclitaxel/Carboplatin Induction (N=408) | Consolidation (Gemcitabine to Paclitaxel) (N=169) | Consolidation (Paclitaxel to Paclitaxel) (N=183) | Crossover (Paclitaxel to Gemcitabine) (N=78) | Crossover (Gemcitabine to Paclitaxel) (N=77)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5) | 9 (11) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (7) | 5 (6) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal infarction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (16) | 8 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retroperitoneum cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (13) | 9 (10) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (10) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Sensation of pressure (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchopneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central line infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected cyst (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pneumonia primary atypical (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis septic (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 6 (9) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug administration error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Absolute neutrophil count/absolute granulocyte count (Investigations) | 21 (24) | 14 (16) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemoglobin (Investigations) | 24 (28) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Platelet count (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelets (Investigations) | 43 (53) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cells (Investigations) | 10 (12) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 6 (6) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemic coma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematologic (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The adverse event term and organ system were not coded via MedDRA. The organ system was provide as a requirement to release the record.
Infection/febrile neutropenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — The adverse event term and organ system were not coded via MedDRA. The organ system was provide as a requirement to release the record.
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Costovertebral angle tenderness (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal infarct (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract disorder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain management (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine/Carboplatin Induction (N=412) | Paclitaxel/Carboplatin Induction (N=408) | Consolidation (Gemcitabine to Paclitaxel) (N=169) | Consolidation (Paclitaxel to Paclitaxel) (N=183) | Crossover (Paclitaxel to Gemcitabine) (N=78) | Crossover (Gemcitabine to Paclitaxel) (N=77)
Lymphopenia (Blood and lymphatic system disorders) | 9 (25) | 10 (25) | 2 (4) | 4 (9) | 4 (10) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 22 (68) | 8 (12) | 1 (4) | 1 (7) | 4 (4) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 18 (31) | 22 (39) | 8 (26) | 14 (39) | 0 (0) | 2 (8)
Vision blurred (Eye disorders) | 15 (26) | 26 (50) | 9 (26) | 15 (33) | 3 (6) | 2 (3)
Visual disturbance (Eye disorders) | 5 (5) | 11 (15) | 8 (15) | 8 (23) | 3 (5) | 4 (9)
Abdominal distension (Gastrointestinal disorders) | 21 (32) | 11 (16) | 9 (24) | 13 (18) | 5 (12) | 5 (10)
Abdominal pain (Gastrointestinal disorders) | 88 (168) | 92 (148) | 29 (76) | 32 (68) | 14 (26) | 16 (30)
Abdominal pain upper (Gastrointestinal disorders) | 21 (27) | 16 (24) | 8 (13) | 7 (10) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 173 (400) | 170 (391) | 54 (154) | 62 (178) | 31 (66) | 25 (60)
Diarrhoea (Gastrointestinal disorders) | 83 (145) | 97 (187) | 43 (107) | 43 (111) | 12 (17) | 9 (19)
Dyspepsia (Gastrointestinal disorders) | 16 (21) | 17 (26) | 9 (24) | 14 (20) | 3 (6) | 5 (6)
Nausea (Gastrointestinal disorders) | 213 (504) | 205 (506) | 67 (191) | 46 (110) | 32 (67) | 21 (48)
Stomatitis (Gastrointestinal disorders) | 25 (33) | 23 (40) | 11 (18) | 8 (24) | 0 (0) | 3 (7)
Vomiting (Gastrointestinal disorders) | 95 (146) | 95 (154) | 19 (24) | 12 (20) | 14 (22) | 9 (20)
Asthenia (General disorders) | 28 (39) | 34 (41) | 7 (12) | 8 (15) | 3 (3) | 2 (2)
Fatigue (General disorders) | 281 (948) | 279 (912) | 108 (531) | 119 (558) | 56 (217) | 40 (160)
Oedema (General disorders) | 20 (31) | 8 (13) | 3 (5) | 8 (18) | 5 (7) | 1 (1)
Oedema peripheral (General disorders) | 46 (84) | 33 (53) | 18 (50) | 21 (64) | 5 (12) | 6 (8)
Pain (General disorders) | 25 (31) | 38 (59) | 36 (76) | 26 (43) | 8 (12) | 4 (6)
Pyrexia (General disorders) | 34 (47) | 19 (24) | 4 (4) | 6 (8) | 9 (10) | 4 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 5 (7) | 5 (7) | 6 (6) | 4 (4) | 0 (0)
Sinusitis (Infections and infestations) | 6 (6) | 13 (18) | 3 (3) | 10 (14) | 7 (8) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 12 (12) | 6 (8) | 7 (10) | 12 (13) | 4 (5) | 0 (0)
Urinary tract infection (Infections and infestations) | 28 (31) | 31 (41) | 10 (15) | 14 (19) | 4 (4) | 4 (5)
Contusion (Injury, poisoning and procedural complications) | 31 (48) | 15 (28) | 9 (12) | 6 (19) | 0 (0) | 1 (2)
Alanine aminotransferase (Investigations) | 24 (53) | 19 (33) | 4 (6) | 7 (21) | 5 (12) | 1 (3)
Alanine aminotransferase increased (Investigations) | 64 (120) | 27 (46) | 10 (27) | 10 (17) | 11 (20) | 2 (10)
Anc/agc (Investigations) | 378 (1638) | 361 (1531) | 88 (314) | 93 (325) | 68 (246) | 47 (173)
Aspartate aminotransferase increased (Investigations) | 58 (100) | 21 (36) | 10 (21) | 13 (23) | 12 (19) | 3 (8)
Blood albumin decreased (Investigations) | 18 (39) | 17 (36) | 2 (2) | 3 (4) | 4 (7) | 1 (1)
Blood alkaline phosphatase (Investigations) | 23 (51) | 20 (32) | 6 (19) | 7 (12) | 3 (7) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 52 (103) | 37 (68) | 13 (33) | 8 (38) | 8 (11) | 7 (12)
Blood glucose (Investigations) | 11 (18) | 22 (32) | 12 (17) | 10 (46) | 0 (0) | 4 (10)
Blood glucose increased (Investigations) | 46 (93) | 50 (108) | 26 (79) | 21 (55) | 10 (13) | 5 (18)
Blood sodium decreased (Investigations) | 14 (28) | 23 (41) | 5 (7) | 7 (9) | 5 (7) | 1 (2)
Blood urea increased (Investigations) | 19 (39) | 18 (28) | 22 (53) | 7 (20) | 3 (4) | 4 (21)
Carbon dioxide increased (Investigations) | 18 (41) | 8 (11) | 12 (33) | 6 (11) | 4 (5) | 2 (4)
Haematocrit (Investigations) | 24 (42) | 17 (33) | 1 (3) | 7 (12) | 1 (9) | 1 (1)
Hemoglobin (Investigations) | 385 (1830) | 352 (1436) | 83 (338) | 103 (375) | 66 (270) | 54 (201)
Hepatic enzyme increased (Investigations) | 5 (8) | 1 (1) | 6 (9) | 2 (2) | 5 (8) | 0 (0)
Liver function test abnormal (Investigations) | 16 (19) | 9 (13) | 2 (12) | 1 (1) | 5 (11) | 2 (3)
Platelets (Investigations) | 379 (1550) | 233 (631) | 36 (110) | 23 (72) | 61 (216) | 16 (31)
Protein total decreased (Investigations) | 9 (10) | 15 (20) | 7 (17) | 1 (1) | 5 (6) | 3 (3)
White blood cells (Investigations) | 380 (1714) | 350 (1507) | 88 (423) | 101 (442) | 68 (247) | 49 (208)
Weight decreased (Investigations) | 37 (67) | 31 (45) | 6 (10) | 6 (7) | 1 (1) | 3 (5)
Weight increased (Investigations) | 24 (60) | 15 (33) | 26 (100) | 31 (88) | 7 (16) | 5 (25)
Anorexia (Metabolism and nutrition disorders) | 49 (82) | 57 (99) | 13 (22) | 5 (8) | 7 (15) | 8 (25)
Hyperglycaemia (Metabolism and nutrition disorders) | 45 (111) | 72 (158) | 36 (150) | 42 (152) | 10 (23) | 16 (53)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 17 (35) | 11 (18) | 0 (0) | 0 (0) | 2 (7) | 5 (6)
Hypocalcaemia (Metabolism and nutrition disorders) | 14 (29) | 8 (12) | 2 (2) | 3 (3) | 3 (3) | 4 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 29 (47) | 20 (29) | 6 (13) | 11 (18) | 2 (3) | 8 (13)
Hyponatraemia (Metabolism and nutrition disorders) | 14 (19) | 14 (24) | 6 (9) | 8 (15) | 0 (0) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 48 (86) | 108 (247) | 66 (192) | 53 (149) | 16 (32) | 25 (62)
Arthritis (Musculoskeletal and connective tissue disorders) | 8 (16) | 4 (6) | 4 (10) | 10 (33) | 2 (6) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 47 (72) | 42 (81) | 19 (37) | 30 (76) | 9 (12) | 8 (12)
Bone pain (Musculoskeletal and connective tissue disorders) | 14 (22) | 33 (45) | 16 (38) | 8 (15) | 1 (1) | 6 (9)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 15 (30) | 26 (46) | 8 (22) | 18 (69) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 25 (41) | 55 (97) | 37 (91) | 25 (53) | 8 (17) | 8 (13)
Myalgia (Musculoskeletal and connective tissue disorders) | 36 (62) | 100 (220) | 44 (130) | 38 (103) | 10 (23) | 17 (40)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (45) | 49 (75) | 18 (45) | 18 (62) | 8 (8) | 6 (6)
Dizziness (Nervous system disorders) | 44 (65) | 34 (52) | 11 (22) | 14 (18) | 6 (10) | 5 (9)
Headache (Nervous system disorders) | 40 (82) | 39 (75) | 20 (41) | 15 (28) | 4 (7) | 6 (14)
Hypoaesthesia (Nervous system disorders) | 25 (36) | 53 (93) | 29 (70) | 33 (103) | 5 (14) | 12 (32)
Neuropathy (Nervous system disorders) | 15 (28) | 65 (140) | 39 (122) | 51 (183) | 7 (20) | 19 (64)
Neuropathy peripheral (Nervous system disorders) | 22 (58) | 99 (190) | 62 (207) | 68 (211) | 17 (39) | 23 (60)
Paraesthesia (Nervous system disorders) | 28 (42) | 88 (191) | 38 (94) | 42 (165) | 15 (27) | 9 (19)
Peripheral sensory neuropathy (Nervous system disorders) | 20 (42) | 61 (162) | 26 (91) | 43 (186) | 9 (22) | 11 (48)
Neurology (Nervous system disorders) | 2 (2) | 10 (17) | 3 (4) | 7 (28) | 1 (1) | 5 (20) — The adverse event term and organ system were not coded via MedDRA. The organ system was provide as a requirement to release the record.
Pain (Nervous system disorders) | 6 (7) | 7 (9) | 1 (1) | 3 (4) | 1 (1) | 5 (15) — The adverse event term and organ system were not coded via MedDRA. The organ system was provide as a requirement to release the record.
Anxiety (Psychiatric disorders) | 32 (63) | 35 (50) | 19 (38) | 15 (35) | 4 (5) | 8 (11)
Depression (Psychiatric disorders) | 47 (92) | 50 (100) | 27 (75) | 36 (132) | 3 (3) | 10 (33)
Insomnia (Psychiatric disorders) | 42 (92) | 73 (150) | 32 (99) | 23 (77) | 9 (12) | 7 (9)
Dysuria (Renal and urinary disorders) | 19 (25) | 21 (26) | 6 (7) | 9 (11) | 3 (3) | 5 (7)
Pollakiuria (Renal and urinary disorders) | 18 (32) | 22 (38) | 7 (9) | 4 (4) | 3 (4) | 3 (6)
Stress urinary incontinence (Renal and urinary disorders) | 3 (6) | 8 (12) | 4 (13) | 10 (34) | 0 (0) | 1 (3)
Urinary incontinence (Renal and urinary disorders) | 7 (13) | 22 (46) | 9 (20) | 7 (24) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 37 (57) | 29 (45) | 22 (49) | 23 (48) | 10 (24) | 5 (21)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 (83) | 67 (99) | 19 (40) | 23 (61) | 11 (14) | 8 (9)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 31 (55) | 20 (27) | 9 (20) | 13 (31) | 4 (15) | 4 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 37 (53) | 13 (22) | 5 (6) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 94 (260) | 249 (917) | 102 (600) | 94 (469) | 42 (117) | 49 (251)
Hypotrichosis (Skin and subcutaneous tissue disorders) | 24 (73) | 9 (12) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (32) | 20 (33) | 10 (18) | 8 (14) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 42 (59) | 42 (68) | 30 (50) | 25 (48) | 8 (9) | 8 (12)
Flushing (Vascular disorders) | 6 (9) | 11 (22) | 10 (14) | 8 (34) | 1 (4) | 1 (2)
Hot flush (Vascular disorders) | 38 (99) | 60 (145) | 35 (132) | 38 (172) | 11 (31) | 6 (22)

LIMITATIONS AND CAVEATS:
Trial was designed with overall survival as primary endpoint. Enrollment was slower than expected. After 4 years, 919 patients were randomized and in August 2006, protocol was amended: primary endpoint was changed to progression free survival (PFS).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days